CLINICAL TRIAL: NCT06348537
Title: Therapeutic Potential of Olive Polyphenols in Fibromyalgia Management
Brief Title: Effects of Olive Polyphenols in Fibromyalgia Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Granada (Other)
Collaborators: Solvitae Medical, S.L (Unknown); University of Jaén (Other)
Responsible Party: Principal Investigator, ALMA RUS MARTÍNEZ, PhD, Universidad de Granada
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Polyphenol-Fibromyalgia
Record Dates: First submitted 2024-03-21; First posted 2024-04-04 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-03

CONDITIONS: Fibromyalgia
Keywords: olive polyphenol; Oxidative stress; Inflammation; coagulation; pain; proteomics
MeSH Terms: conditions — Fibromyalgia; Inflammation; Thrombosis; Pain

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): Group 1: consisting of 20 patients diagnosed with FM, who received a daily dose of 3 capsules (2 in the morning and 1 in the evening) of Mygrium® during 60 days.
  Interventions: Dietary Supplement: Olive Polyphenols
- Group 2 (Placebo Comparator): Group 2: 20 patients diagnosed with FM, who received a daily dose of 3 capsules (2 in the morning and 1 in the evening) of a placebo (maltodextrins) during 60 days. This intervention group served as a control.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Olive Polyphenols — Patients with fibromyalgia of Group 1 will consume Olive Polyphenols daily during 60 days.
  Arms: Group 1
Dietary Supplement: Placebo — Patients with fibromyalgia of Group 2 will consume a placebo daily during 60 days.
  Arms: Group 2

SUMMARY:
To study the effects of a nutritional intervention with an olive (poly)phenol preparation in female patients with FM.

DETAILED DESCRIPTION:
This work has studied the effects of a nutritional intervention with an olive (poly)phenol preparation in female patients with FM, analyzing the complete blood count, the biochemical, lipid and coagulation profiles as well as the inflammatory and oxidative statuses in blood samples.

ELIGIBILITY:
Inclusion Criteria:

* Patients to be included in the study must be female over 18 years of age. The patients had to be previously diagnosed with FM according to the criteria of the American College of Rheumatology.

Exclusion Criteria:

* Other chronic diseases: diabetes mellitus, hypertension, cardiovascular disorders, cancer…
* Patients with grade II obesity (body mass index ≥ 35 kg/m2).
* Active smokers.
* Pregnancy.
* Regular treatment with acetylsalicylic acid, estrogen, corticosteroids, antioxidants or lipid-lowering drugs.
* Participation in another research study.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-01-20 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Plasma proteome | It will be carried out on blood samples from the study participants before starting the intervention and at the end. Estimated duration of 3 months
  Proteomic analyses will be performed by liquid nano-chromatography coupled to label-free tandem mass spectrometry (label-free nLC-MS/MS). This technique allows the relative quantification of the abundance of each protein in each sample, making it possible to assess those with differential expression in the different study groups.
Lipid peroxidation | It will be carried out on blood samples from the study participants before starting the intervention and at the end. Estimated duration of 1 month
  Lipid peroxidation is determined by thiobarbituric acid reactive substances (TBARS) method.

SECONDARY OUTCOMES:
Aldolase | It will be carried out on blood samples from the study participants before starting the intervention and at the end. Estimated duration of 1 month
  Aldolase is measured using an AU 5800 analyzer (Beckman Coulter).
C-reactive protein (CRP) | It will be carried out on blood samples from the study participants before starting the intervention and at the end. Estimated duration of 1 month
  C-reactive protein (CRP) ie measured using an AU 5800 analyzer (Beckman Coulter).
Impact of fibromyalgia | It will be carried out on blood samples from the study participants before starting the intervention and at the end. Estimated duration of 20 minutes
  FIQR (Revised Fibromyalgia Impact Questionnaire) will be used to evaluate the functional capacity in daily living activities
Quality of Life | It will be carried out on blood samples from the study participants before starting the intervention and at the end. Estimated duration of 20 minutes
  SF-12 (Quality of Life Questionnaire) is used to assess quality of life.
Red blood cells | It will be carried out on blood samples from the study participants before starting the intervention and at the end. Estimated duration of 1 month
  Red blood cells are measured using a DxH 900 Workcell Automated Hematology Solution (Beckman Coulter).
Haemoglobin | It will be carried out on blood samples from the study participants before starting the intervention and at the end. Estimated duration of 1 month
  Haemoglobin is measured using a DxH 900 Workcell Automated Hematology Solution (Beckman Coulter).
Fibrinogen | It will be carried out on blood samples from the study participants before starting the intervention and at the end. Estimated duration of 1 month
  Fibrinogen is measured using a DxH 900 Workcell Automated Hematology Solution (Beckman Coulter).
Total cholesterol | It will be carried out on blood samples from the study participants before starting the intervention and at the end. Estimated duration of 1 month
  Total cholesterol is measured by a spectrophotometric procedure using an Olympus AU 5400 analyzer (Beckman Coulter).
Cholesterol ratio | It will be carried out on blood samples from the study participants before starting the intervention and at the end. Estimated duration of 1 month
  Cholesterol ratio is measured by a spectrophotometric procedure using an Olympus AU 5400 analyzer (Beckman Coulter).
LDL cholesterol | It will be carried out on blood samples from the study participants before starting the intervention and at the end. Estimated duration of 1 month
  LDL cholesterol is measured by a spectrophotometric procedure using an Olympus AU 5400 analyzer (Beckman Coulter).
Cortisol | It will be carried out on blood samples from the study participants before starting the intervention and at the end. Estimated duration of 1 month
  Cortisol level is determined in serum samples by a fluorescence polarization immunoassay using an AxSYM (Abbott Laboratories, IL, USA).

CONTACTS AND LOCATIONS:
Overall Officials: Mª Luisa del Moral, MD, Principal Investigator — University of Jaén
Locations (1):
- University of Jaén, Jaén, Spain

REFERENCES:
- [Derived] de la Cruz Cazorla S, Blanco S, Rus A, Molina-Ortega FJ, Ocana E, Hernandez R, Visioli F, Moral MLD. Nutraceutical Supplementation as a Potential Non-Drug Treatment for Fibromyalgia: Effects on Lipid Profile, Oxidative Status, and Quality of Life. Int J Mol Sci. 2024 Sep 14;25(18):9935. doi: 10.3390/ijms25189935. PMID 39337423